CLINICAL TRIAL: NCT00452335
Title: A Multi-center, Open-labeled Study of the Safety, Efficacy, and Pharmacokinetics of Lubiprostone in Pediatric Patients With Constipation
Brief Title: Safety and Efficacy of Lubiprostone in Pediatric Patients With Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Sucampo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0211SC-0641
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-07

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lubiprostone 12 mcg QD (Experimental): Children (6-11 years of age) who are at least 12 kg, but less than 24 kg, body weight, and young children (<6 years of age and able to swallow capsules) who are at least 12 kg body weight
  Interventions: Drug: Lubiprostone
- Lubiprostone 12 mcg BID (Experimental): Up to 24 adolescents (12-17 years of age) and all children (6-11 years of age) who are at least 24 kg, but less than 36 kg, body weight
  Interventions: Drug: Lubiprostone
- Lubiprostone 24 mcg BID (Experimental): Adolescents (12-17 years of age)and children (6-11 years of age) who are ≥36 kg body weight
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone — 12 mcg capsule once daily (QD)
  Other Names: Amitiza®
  Arms: Lubiprostone 12 mcg QD
Drug: Lubiprostone — 12 mcg capsule twice daily (BID)
  Other Names: Amitiza®
  Arms: Lubiprostone 12 mcg BID
Drug: Lubiprostone — 24 mcg capsule twice daily (BID)
  Other Names: Amitiza®
  Arms: Lubiprostone 24 mcg BID

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of lubiprostone in a pediatric population with constipation, including the pharmacokinetics of lubiprostone, in a subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 years of age
* Weight of at least 12 kg and capable of swallowing a capsule
* Able to refrain from use of medications known to treat or associated with constipation symptoms
* Stable fiber therapy or ADHD therapy if using such medications
* Patient/Caregiver able to complete daily diary
* Patient able to use recommended rectal and/or oral rescue medications if needed

Exclusion Criteria:

* Constipation is associated with some medical, anatomic, physical, organic, or other condition
* Hirschsprung's Disease or Nonretentive Fecal Incontinence
* Untreated fecal impactions or impactions requiring digital manipulation
* Open gastrointestinal/abdominal surgery or laparoscopic surgery at the investigator discretion
* Organic bowel disorder, mechanical bowel obstruction, pseudo-obstruction, or unexplained weight loss
* Uncontrolled cardiovascular, liver or lung disease, neurologic or psychiatric disorder, other systemic disease, or abnormal laboratory tests at the investigator discretion
* If female, is currently pregnant or nursing, or plans to become pregnant or nurse during the clinical study
* Sexually active males and females must utilize acceptable birth control methods
* Prior use of lubiprostone, Amitiza, SPI-0211, or RU-0211

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2007-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hyman, MD, Principal Investigator — University of Kansas Medical Center
Locations (19):
- United States (19):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Center for Children's Digestive Health, Park Ridge, Illinois
  - University of Illinois at Peoria, Peoria, Illinois
  - University of Illinois at Chicago, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Hospital Boston, Boston, Massachusetts
  - The Center for Human Nutrition, Inc., Omaha, Nebraska
  - AHS Hospital Corporation, Morristown, New Jersey
  - Children's Research Institute, Columbus, Ohio
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - Southeastern Clinical Research, Chattanooga, Tennessee
  - Jackson Clinic, Jackson, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 127 participants were randomized to study treatment, however only 124 participants received study drug
Groups:
- 12 mcg QD: Children (6-11 years of age) who are at least 12 kg, but less than 24 kg, body weight, and young children (<6 years of age and able to swallow capsules) who are at least 12 kg body weight
- 12 mcg BID: Up to 24 adolescents (12-17 years of age) and all children (6-11 years of age) who are at least 24 kg, but less than 36 kg, body weight
- 24 mcg BID: Adolescents (12-17 years of age)and children (6-11 years of age) who are ≥36 kg body weight
Period: Overall Study
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID
Started | 27 | 65 | 32
Completed | 25 | 61 | 23
Not Completed | 2 | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID | Total
Number analyzed (Participants) | 27 | 65 | 32 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 65 | 32 | 124
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (1.67) | 10.3 (2.78) | 13.9 (3.00) | 10.2 (3.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 24 | 23 | 59
  Male | 15 | 41 | 9 | 65
Region of Enrollment [Number; unit: participants]
  United States | 27 | 65 | 32 | 124

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Spontaneous Bowel Movements
Description: Gathered as part of the daily electronic diary questions.
Time Frame: Week 1
Population: ITT population
Measure: Mean (Standard Deviation); unit: spontaneous bowel movements per week
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID
Number analyzed (Participants) | 27 | 65 | 31
spontaneous bowel movements per week | 2.47 (2.68) | 3.02 (2.17) | 3.84 (2.51)

2. Secondary Outcome: Frequency of Spontaneous Bowel Movements
Description: Gathered as part of the daily electronic diary questions.
Time Frame: Weeks 2, 3, and 4
Population: ITT Population
Measure: Mean (Standard Deviation); unit: spontaneous bowel movements per week
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID
Number analyzed (Participants) | 27 | 65 | 31
spontaneous bowel movements per week
  Week 2 | 2.79 (2.278) | 2.59 (2.316) | 3.51 (1.897)
  Week 3 | 2.64 (2.210) | 2.60 (2.006) | 3.58 (2.422)
  Week 4 | 2.85 (2.130) | 2.68 (2.258) | 2.99 (1.827)

3. Secondary Outcome: Frequency of Fecal Incontinence
Description: As part of the daily diary, patients were asked to report the number of fecal incontinence episodes per day.
Time Frame: Weekly, up to 4 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: episodes of fecal incontinence per day
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID
Number analyzed (Participants) | 27 | 65 | 31
episodes of fecal incontinence per day
  Week 1 | 0.53 (1.141) | 0.22 (0.489) | 0.03 (0.089)
  Week 2 | 0.37 (0.768) | 0.21 (0.446) | 0.05 (0.148)
  Week 3 | 0.40 (0.989) | 0.16 (0.336) | 0.01 (0.060)
  Week 4 | 0.48 (1.168) | 0.17 (0.457) | 0.02 (0.074)

4. Secondary Outcome: Straining Associated With SBMs
Description: Bowel straining assessed based on the following scale: 0 = no straining, 1 = mild straining, 2 = moderate straining, 3 = severe straining, and 4 = very severe straining.
Time Frame: Weekly, up to 4 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 24 Mch BID: Adolescents (12-17 years of age)and children (6-11 years of age) who are ≥36 kg body weight
Arm/Group | 12 mcg QD | 12 mcg BID | 24 Mch BID
Number analyzed (Participants) | 27 | 65 | 31
units on a scale
  Week 1 | 1.70 (1.074) | 1.34 (1.001) | 1.44 (0.890)
  Week 2 | 1.02 (1.010) | 1.22 (0.868) | 1.30 (1.003)
  Week 3 | 1.11 (0.857) | 1.11 (0.809) | 1.16 (1.130)
  Week 4 | 1.03 (0.887) | 1.31 (1.096) | 0.97 (1.089)

5. Secondary Outcome: Stool Consistency of SBMs
Description: Stool consistency was captured using the Bristol Stool Form Scale: 1 = Separate hard lumps like nuts, 2 = Sausage shaped but lumpy, 3 = Like a sausage but with cracks on surface, 4 = Like a sausage or snake, smooth and soft, 5 = Soft blobs with clear-cut edges, 6 = Fluffy pieces with ragged edges, a mushy stool, and 7 = Watery, no solid pieces.
Time Frame: Weekly, up to 4 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID
Number analyzed (Participants) | 27 | 65 | 31
units on a scale
  Week 1 | 2.87 (1.197) | 3.20 (1.168) | 3.14 (1.249)
  Week 2 | 3.09 (1.078) | 2.90 (1.198) | 3.22 (1.394)
  Week 3 | 2.93 (0.796) | 3.31 (1.121) | 3.59 (1.168)
  Week 4 | 3.20 (0.904) | 2.96 (1.160) | 4.01 (1.631)

6. Secondary Outcome: Abdominal Bloating
Description: Abdominal bloating was assessed based on the following scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe.
Time Frame: Weekly, up to 4 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID
Number analyzed (Participants) | 27 | 65 | 31
units on a scale
  Week 1 | 1.16 (0.800) | 1.39 (1.150) | 1.79 (0.876)
  Week 2 | 1.08 (0.929) | 1.12 (1.027) | 1.16 (0.987)
  Week 3 | 0.82 (1.006) | 1.00 (0.937) | 1.08 (1.018)
  Week 4 | 0.96 (1.065) | 1.04 (0.865) | 1.05 (0.950)

7. Secondary Outcome: Abdominal Discomfort
Description: Abdominal discomfort was assessed based on the following scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe.
Time Frame: Weekly, up to 4 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 12 mcg BID | 12 mcg QD | 24 mcg BID
Number analyzed (Participants) | 27 | 65 | 31
units on a scale
  Week 1 | 0.84 (0.800) | 1.16 (1.134) | 1.43 (1.289)
  Week 2 | 1.08 (0.929) | 0.93 (0.918) | 1.20 (1.080)
  Week 3 | 0.82 (0.795) | 0.90 (0.892) | 1.17 (1.204)
  Week 4 | 0.87 (0.869) | 1.05 (0.915) | 1.14 (1.125)

8. Secondary Outcome: Pain Associated With SBMs
Description: Pain associated with SBMs was assessed based on the following scale: 0 = no pain, 1 = mild pain, 2 = moderate pain, 3 = severe pain, and 4 = very severe pain.
Time Frame: Weekly, up to 4 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID
Number analyzed (Participants) | 27 | 65 | 31
units on a scale
  Week 1 | 1.56 (1.051) | 1.13 (0.970) | 1.14 (0.873)
  Week 2 | 0.72 (1.009) | 1.06 (0.758) | 1.10 (1.073)
  Week 3 | 0.88 (0.929) | 0.91 (0.915) | 1.01 (1.089)
  Week 4 | 0.82 (0.978) | 1.07 (1.047) | 1.07 (1.298)

9. Secondary Outcome: Constipation Severity
Description: Constipation severity was assessed based on the following scale 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe.
Time Frame: Weekly, up to 4 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID
Number analyzed (Participants) | 27 | 65 | 31
units on a scale
  Week 1 | 1.92 (1.038) | 1.69 (0.951) | 1.79 (0.917)
  Week 2 | 1.46 (0.977) | 1.43 (0.945) | 1.40 (0.816)
  Week 3 | 1.59 (0.908) | 1.36 (1.055) | 1.38 (0.875)
  Week 4 | 1.43 (1.121) | 1.28 (1.031) | 1.59 (1.054)

10. Secondary Outcome: Treatment Effectiveness
Description: Treatment effectiveness was assessed with the following scale: 0 = not at all effective, 1 = a little bit effective, 2 = moderately effective, 3 = quite a bit effective, and 4 = extremely effective.
Time Frame: Weekly, up to 4 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID
Number analyzed (Participants) | 27 | 65 | 31
units on a scale
  Week 1 | 1.2 (1.30) | 1.6 (1.27) | 1.7 (0.86)
  Week 2 | 1.6 (1.28) | 1.7 (1.24) | 2.0 (1.17)
  Week 3 | 1.9 (1.51) | 1.8 (1.31) | 1.8 (1.24)
  Week 4 | 2.0 (1.43) | 1.8 (1.22) | 1.9 (1.10)

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs: up to 4 weeks plus 7 days (from time of first dose to 7 days post-treatment)
Arm/Group | 12 mcg QD | 12 mcg BID | 24 mcg BID
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/65 | 0/32
Other Adverse Events (participants affected / at risk) | 5/27 | 23/65 | 14/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 12 mcg QD (N=27) | 12 mcg BID (N=65) | 24 mcg BID (N=32)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 12 mcg QD (N=27) | 12 mcg BID (N=65) | 24 mcg BID (N=32)
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 3
Nausea (Gastrointestinal disorders) | 1 | 12 | 10
Vomiting (Gastrointestinal disorders) | 4 | 6 | 5
Headache (Nervous system disorders) | 0 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days